CLINICAL TRIAL: NCT04916379
Title: Effect of Momordica Charantia Administration on Anthropometric Indicators in Patients With Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Marisol Cortez Navarrete, Principal investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCHOB
Record Dates: First submitted 2021-06-02; First posted 2021-06-07 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: Momordica charantia; Bitter melon; Obesity
MeSH Terms: conditions — Obesity | interventions — bitter melon extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Momordica charantia (Experimental): Two 500 mg capsules of Momordica charantia twice daily before breakfast and dinner for 12 weeks
  Interventions: Dietary Supplement: Momordica charantia
- Placebo (Placebo Comparator): Two 500 mg capsules of calcined magnesia twice daily before breakfast and dinner for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Momordica charantia — Momordica Charantia: 2000 mg per day for 12 weeks
  Other Names: Bitter melon
  Arms: Momordica charantia
Other: Placebo — Placebo: 2000 mg per day for 12 weeks
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
Momordica charantia has shown to exert anti-obesity effects through numerous mechanisms of action described in preclinical studies. Important reductions in body weight and other anthropometric indicators have been reported in clinical trials. However, these beneficial effects of Momordica charantia on obesity have been observed mainly in type 2 diabetes mellitus patients. The purpose of this study is to evaluate the effect of Momordica charantia administration on anthropometric indicators in patients with obesity.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo controlled clinical trial is carried out in 24 patients with obesity according to the body mass index.

Patients are assigned to two different arms: one group receives Momordica charantia, 2 capsules with 500 mg twice daily before breakfast and dinner for 12 weeks or placebo, under the same scheme of treatment.

Body weight, body mass index, waist circumference, body fat percentage and other clinical and laboratory parameters are evaluated.

This protocol is approved by a local ethics committee and written informed consent will be obtained from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity type I according to body mass index (IMC: 30.0 - 34.9 kg/m2)
* Body weight without variations above or under 5% in the last three months before entering the study
* Fasting plasma glucose: <126 mg/dL
* Total cholesterol: <240 mg/dL
* Triglycerides: <400 mg/dL
* Women in childbearing years must have a contraceptive method
* Letter of consent and release signed by each patient

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Known uncontrolled renal, hepatic, cardiovascular or thyroid disease
* Physical impossibility for taking pills
* Known hypersensibility to the Momordica charantia or placebo

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline body mass index (BMI) at 12 weeks | 12 weeks
  BMI is calculated at baseline and after 12 weeks with the Quetelet index formula
Change from baseline body weight (BW) at 12 weeks | 12 weeks
  BW is evaluated at baseline and after 12 weeks with an electric bioimpedance digital scale (Model TBF-300 A; Tanita Corporation of America Inc., Arlington Heights, IL)
Change from baseline fat mass at 12 weeks | 12 weeks
  Fat mass is measured at baseline and after 12 weeks with an electric bioimpedance digital scale (Model TBF-300 A; Tanita Corporation of America Inc., Arlington Heights, IL)
Change from baseline waist circumference (WC) at 12 weeks | 12 weeks
  WC is evaluated at baseline and after 12 weeks with a flexible tape in the midpoint between the lowest rib and the iliac crest

SECONDARY OUTCOMES:
Change from baseline fasting plasma glucose (FPG) at 12 weeks | 12 weeks
  FPG is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline total cholesterol at 12 weeks | 12 weeks
  Total cholesterol is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline triglycerides at 12 weeks | 12 weeks
  Triglycerides are evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline high density lipoprotein cholesterol (HDL-c) at 12 weeks | 12 weeks
  HDL-c is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline low density lipoprotein cholesterol (LDL-c) at 12 weeks | 12 weeks
  LDL-c is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline very low density lipoprotein (VLDL) at 12 weeks | 12 weeks
  VLDL is calculated at baseline and after 12 weeks as triglycerides/5
Change from baseline creatinine at 12 weeks | 12 weeks
  Creatinine is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline uric acid at 12 weeks | 12 weeks
  Uric acid is evaluated at baseline and after 12 weeks with enzymatic-colorimetric techniques
Change from baseline alanine aminotransferase (ALT) at 12 weeks | 12 weeks
  ALT is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline aspartate aminotransferase (AST) at 12 weeks | 12 weeks
  AST is evaluated at baseline and after 12 weeks with enzymatic/colorimetric techniques
Change from baseline systolic blood pressure at 12 weeks | 12 weeks
  Systolic blood pressure is measured at baseline and after 12 weeks with a digital sphygmomanometer
Change from baseline diastolic blood pressure at 12 weeks | 12 weeks
  Diastolic blood pressure is measured at baseline and after 12 weeks with a digital sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Cortez Navarrete, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Cortez-Navarrete M, Mendez-Del Villar M, Martinez-Abundis E, Lopez-Murillo LD, Escobedo-Gutierrez MJ, Rosales-Rivera LY, Perez-Rubio KG. Effect of Momordica charantia Administration on Anthropometric Measures and Metabolic Profile in Patients with Obesity: A Pilot Clinical Trial. J Med Food. 2022 Jun;25(6):645-651. doi: 10.1089/jmf.2021.0164. Epub 2022 May 4. PMID 35507955